CLINICAL TRIAL: NCT05172453
Title: A Real World, Multi-center Study on Mother-to-child Transmission of Hepatitis B Virus in China
Brief Title: Mother-to-child Transmission of HBV in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Chinese Foundation for Hepatitis Prevention and Control (Unknown); Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jinlin Hou, Professor & Director, Nanfang Hospital, Southern Medical University
Other Study IDs: shield project 02
Record Dates: First submitted 2021-12-01; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B, Chronic; Mother to Child Transmission
Keywords: hepatitis B; mother-to-child transmission
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nationwide hospital-based cohort: HBV-infected mother-infant pairs have been followed from registry to post vaccination serological test (PVST) in hospitals nationwide.
  Interventions: Other: comprehensive management algorithm for preventing mother-to-child transmission of HBV
- Community-based cohort: HBV-infected mother-infant pairs have been followed from registry to post vaccination serological test (PVST) in Bao' an district, Shenzhen
  Interventions: Other: comprehensive management algorithm for preventing mother-to-child transmission of HBV

INTERVENTIONS:
Other: comprehensive management algorithm for preventing mother-to-child transmission of HBV — To standardize the clinical management of preventing MTCT of HBV and reduce incidences of MTCT, the Chinese Foundation for Hepatitis Prevention and Control (CFHPC) organized experts to compile the "Management algorithm for prevention of mother-to-child transmission of hepatitis B virus" based on the latest research progress and recently published guidelines, which includes 10 steps of pregnancy management and postpartum follow-up, among which screening, antiviral treatment, and infant immunization are its core contents.

SUMMARY:
In order to evaluate the feasibility of eliminating mother-to-child transmission (MTCT) of hepatitis B virus (HBV) by 2030, a multi-center, prospective cohorts study was conducted to investigate MTCT of HBV in China.

DETAILED DESCRIPTION:
A prospective, multicenter study of pregnant women with HBV infection was conducted from July 2015 up to now in a real world setting in the Shield Project stage Ⅱ. Inclusion criteria was any pregnant women with chronic HBV infection. Pregnant women were excluded if they had a positive serologic test for human immunodeficiency virus or hepatitis C virus or any co-morbidity that might reduce compliance or if they were unable or unwilling to use the mobile health application-Shield APP. Enrolled mothers and infants were prospectively followed until infant post-vaccination serologic testing (PVST) was performed at 7-12 months of age.

Demographic data, antiviral treatment history, pregnancy and labour history, co-morbidity, HBV serologic marker tests, HBV DNA tests, liver function tests, mode of delivery, neonatal characteristics (height, weight, head circumference, Apgar score and any major birth defect), breastfeeding and PVST for infants at 7-12 months of age were collected.

A mobile health application called "SHIELD" was developed and used in the Shield Project stage Ⅱ to collect data and provide support for communication between mothers and their doctors. All laboratory test reports, questionnaires and other relevant information was uploaded into SHIELD. Participants could consult with their doctors via SHIELD during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with chronic HBV infection.

Exclusion Criteria:

* positive serologic test for human immunodeficiency virus or hepatitis C virus;
* any co-morbidity that might reduce compliance;
* unable or unwilling to use the mobile health application-Shield APP

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — To investigate mother-to-child transmission, only pregnant women were included.
Study Population: Pregnant women with HBV infection in more than 100 hospitals covering 31 regions in China from Jul 2015 to Jun 2021 were enrolled as hospital-based cohort. In addition, pregnant women with HBV infection in Baoan district of Shenzhen, China from Jun 2017 to Dec 2019 were enrolled as community-based cohort.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of mother-to-child transmission of HBV | 5 years
  compare rate of mother-to-child transmission of HBV among children born to mothers with and without antiviral therapy during pregnancy
rate of birth defect | 5 years
  compare rate of birth defect among children born to mothers with and without antiviral therapy during pregnancy

SECONDARY OUTCOMES:
change of HBV DNA level in mothers with antiviral therapy from baseline to withdrawal of antiviral drugs | from enrollment to delivery, assessed up to 40 weeks
  compare HBV DNA levels of mothers with antiviral therapy at baseline and after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (15):
- China (15):
  - Jinlin Hou, Guangzhou, Guangdong
  - 302 military hospital of China, Beijing
  - Beijing YouAn Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Jilin University, Changchun
  - The First People's Hospital of Foshan, Foshan
  - Fifth Affiliated Hospital of Southern Medical University, Guangzhou
  - Guangdong Maternal and Child Care Hospital, Guangzhou
  - Guangzhou No. 8 People's Hospital, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Xixi Hospital of Hangzhou, Hangzhou
  - Third Hospital of Jiujiang, Jiujiang
  - Second Hospital of Nanjing, Nanjing
  - Shanghai Public Health Clinical Center, Shanghai
  - Shenzhen Baoan Maternal and Child Care Hospital, Shenzhen
  - The Third People's Hospital of Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there is no such plan to make IPD available to other researchers.